CLINICAL TRIAL: NCT05113693
Title: A Randomized, Open-label, Single Dose, Crossover Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-393 in Healthy Volunteers Under Fed Conditions
Brief Title: Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-393
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A98_05BE2118
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lobeglitazone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Period 1 - A single dose of 4 tablets(CKD-501 1T, D759 1T, H053 2T) under fed condition.
  Period 2 - A single dose of 2 tablets(CKD-393 2T) under fed condition.
  Interventions: Drug: CKD-393; Drug: CKD-501, D759, H053
- 2 (Experimental): Period 1 - A single dose of 2 tablets(CKD-393 2T) under fed condition.
  Period 2 - A single dose of 4 tablets(CKD-501 1T, D759 1T, H053 2T) under fed condition.
  Interventions: Drug: CKD-393; Drug: CKD-501, D759, H053

INTERVENTIONS:
Drug: CKD-393 — QD, PO
Drug: CKD-501, D759, H053 — QD, PO

SUMMARY:
Objective

- Evaluation of the pharmacokinetic properties and safety of CKD-393 0.25/50/750 mg oral administration in healthy adults under fed condition.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged 19 ≤ ~ < 55-year-old.
2. Weight ≥55kg (man) or 45kg (woman), with calculated body mass index (BMI) of 17.5 ≤ ~ < 30.5 kg/m2.
3. Those who have no congenital diseases or chronic diseases within 3 years and have no abnormal symptoms or findings.
4. Those who are eligible for clinical trials based on laboratory (hematology, blood chemistry, serology, urology) and 12-lead ECG results at screening.
5. Those who voluntarily decide to participate and agree to comply with the cautions after fully understand the detailed description of this clinical trial.
6. Those who agree to contraception until the 1 month after last administration of clinical trial drugs.
7. Those who have the ability and willingness to participate during the entire clinical trail.

Exclusion Criteria:

1. Those who have clinically significant disease or medical history of heart failure, Hepatopathy, Type 1 Diabetes, Diabetic ketoacidosis, Edema, Renal dysfunction, galactose intolerance, glucose-galactose malabsorption. And Those who receive intravenous administration of radioactive iodine contrast agents (for intravenous urography, venous cholangiography, angiography, computed tomography using contrast agents, etc.) during clinical trial.
2. Those who have past medical history of gastrointestinal disorder (Crohn's disease, ulcerative colitis, etc. except simple appendectomy or hernia surgery), which affect the absorption of investigational drug.
3. Those who have the test results written below

   * AST, ALT > 2 times higher than upper normal level
4. Those who exceeding an alcohol consumption criteria(210g/week) within 6 months before the first administration of investigational drug.

   * Beer 1 glass(250ml, Alcohol contents 5%) = 10g
   * Soju 1 glass(50ml, Alcohol contents 20%) = 8g
   * Wine 1 glass(125ml, Alcohol contents 12%) = 12g
5. Those who exceeding smoking criteria(20 cigarettes/day) within 6 months before the first administration of investigational drug.
6. Those who received investigational durg by participating in other clinical trial within 6 months before the first administration of investigational drug.
7. Those who have vital sign written below

   * systolic blood pressure ≥140 mmHg or < 90 mmHg
   * diastolic blood pressure ≥ 90 mmHg or < 60 mmHg
8. Those who have a drug or alcohol abuse history within 1 year before the first administration of investigational drug.
9. Those who take barbiturate and related (causing induction or inhibition. of metabolism) drug within 30 days before the first administration of investigational drug.
10. Those who received Ethical-the-counter (ETC) drugs or Over-the-counter (OTC) drugs within 10 days before the first administration of investigational drug.
11. Those who donated whole blood within 2 months or apheresis within 1 month before the first administration of investigational drug.
12. Those who severe acute/chronic medical or mental condition which can increase the safety risk by administration of investigational drug.
13. Those who have history of hypersensitivity to active pharmaceutical ingredient or additives.
14. Those who are pregnant or breastfeeding.
15. Those who can't ingest a high fat diet.
16. Those who are deemed inappropriate to participate in clinical trial by investigators.

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-501, D759, H053 | Pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hour
  AUCt: Area under the concentration-time curve from time zero to time
Cmax of CKD-501, D759, H053 | Pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hour
  Cmax: Maximum plasma concentration of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Min Gul Kim, M.D, Ph.D., Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea